CLINICAL TRIAL: NCT04749641
Title: Enhanced Histone H3.3-K27M Neoantigen Vaccine Therapy Against Diffuse Intrinsic Pontine Glioma (ENACTING)- A Phase I Clinical Trial
Brief Title: Neoantigen Vaccine Therapy Against H3.3-K27M Diffuse Intrinsic Pontine Glioma
Acronym: ENACTING
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yang Zhang (Other)
Collaborators: TCRCure Biopharma Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yang Zhang, Department of Neurosurgery, Beijing Tiantan Hospital, Capital Medical University, No.119 South Fourth Ring West Road, Fengtai District, Beijing,100070 P.R.China, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY 2019-126-01
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open surgical biopsy (Experimental): A total of 15 subjects with open surgical biopsy indications will receive microsurgical resection, followed by conformal radiotherapy and administration of the researched vaccine.
  Interventions: Biological: Histone H3.3-K27M Neoantigen Vaccine Therapy
- Stereotactic biopsy (Experimental): A total of 15 subjects without open surgical biopsy indications will receive stereotactic biopsy, followed by conformal radiotherapy and administration of the researched vaccine.
  Interventions: Biological: Histone H3.3-K27M Neoantigen Vaccine Therapy

INTERVENTIONS:
Biological: Histone H3.3-K27M Neoantigen Vaccine Therapy — The researched vaccine, containing H3.3-K27M-targeting neoantigen peptides and poly ICLC, will be administered through subcutaneous injection into DIPG patients after they complete surgical/stereotactic biopsy and conformal radiotherapy. The day of first vaccine injection is defined as D1 (day 1), and then the injections will be administered on D3, D15, Day 29, Day 57, Day 85 and one injection every 8 weeks thereafter. In order to determine the Maximum Tolerated Dose (MTD) of the vaccine, a "6+3" dose escalation design is applied. There are three doses for the vaccine. Dose 1: 0.5mg peptide + Poly ICLC; Dose 2: 1mg peptide + Poly ICLC; Dose 3: 2mg peptide + Poly ICLC.

SUMMARY:
Diffuse intrinsic pontine gliomas (DIPGs), which diffusely occupy the pons of brainstem, are the deadliest primary brain cancer in children. Biopsy for pathology plus radiotherapy remains the current standard-of-care treatment that is minimal effective. Thus, the median overall survival after diagnosis is just 10 months. Recent studies have identified a lysine 27-to-methionine (K27M) somatic mutation at histone H3 variant (H3.3), as a feature mutation in DIPGs. Several preclinical studies have already demonstrated H3.3-K27M as a promising target for immunotherapy. The researched vaccine is a cancer-treatment vaccine containing an H3.3-K27M targeted neoantigen peptide, that can be taken up by antigen-presenting cells (APCs). APCs can present the peptide with the major histocompatibility complex (MHC) molecules on cell surface, thereby activating neoantigen-specific T cells and triggering corresponding cytotoxic T cell immune responses to eliminate H3.3-K27M-expressing DIPG cells. The main goal of this study is investigating the safety and preliminary efficacy of the vaccine in treating newly-diagnosed DIPGs when the vaccine is administered in combination with the standard-of-care treatment.

ELIGIBILITY:
Inclusion Criteria:

A. First entry criteria

1. Age ≥ 5 years old;
2. Newly-diagnosed patients with DIPG appearance on MRI image;
3. HLA-A2 subtype;
4. The expected survival time exceeds 24 weeks;
5. The KPS score is greater than 50; B. Second entry criteria

1. The KPS score is greater than 50; 2. DIPG is diagnosed histologically on tumor tissue obtained by biopsy or surgical resection; 3. H3.3K27M mutation is detected on tumor tissue obtained by biopsy or surgical resection ; 4. Adequate organ functions that meet the following criteria: The absolute number of neutrophils: ≥1500/mm3 Platelet count: ≥75000/uL Hemoglobin: ≥80 g/L Creatinine≤1.5×ULN Bilirubin≤1.5×ULN ALT≤3×ULN AST≤3×ULN 5. Ability to comprehend and sign an informed consent form.

Exclusion Criteria:

1. With past medical history of malignant tumors (except being asymptomatic for more than 3 years);
2. History of allergy to chemotherapeutics or radiosensitizers for the treatment of cancer in central nervous system and head/neck;
3. History of allergy to the vaccine and its ingredients;
4. Comorbidity with HIV infection and/or acute phase of hepatitis B/C;
5. Any progressive diseases that hinder participation in the trial;
6. With unstable cardiovascular diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia et.al.;
7. History of uncontrolled mental illnesses;
8. Inability to comprehend or sign informed consent form or abide by the research procedures;
9. Other conditions believed to hinder participation in this trial at investigator' discretion.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Safety of histone H3.3-K27M neoantigen vaccine in treating newly diagnosed DIPGs | All the Adverse events (AEs) were recorded until 24 weeks after the last shot
  AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Rate of the patients who survive for more than one year after surgery/biopsy in all the DIPG patients who receive H3.3-K27M neoantigen vaccine | One year after surgery or biopsy
  One-year survival rate

SECONDARY OUTCOMES:
Maximum Tolerated Dose of H3.3-K27M neoantigen vaccine to treat DIPGs | DLTs were monitored at timepoints of every vaccine shot until the 28th day after the first injection
  ">= Grade 3 " vaccine related AEs are defined as DLTs. In order to determine the Maximum Tolerated Dose (MTD) of the vaccine, a "6+3" dose escalation design is applied.
Rate of the patients who survive for more than two years after surgery/biopsy in all the DIPG patients who receive H3.3-K27M neoantigen vaccine | two years after surgery or biopsy
  two-year survival rate
Median Progression-free survival time of the DIPG patients who receive H3.3-K27M neoantigen vaccine | start 4 weeks after the first shot and every 8 weeks until disease progression
  Progression-free survival time: the time from operation/biopsy to progression (when shows signs or symptoms of the growth or the spreading of a tumor)
Median Overall survival time of the DIPG patients who receive H3.3-K27M neoantigen vaccine | start 4 weeks after the first shot and every 8 weeks until death
  overall survival time: the time from operation/biopsy to death.
Immunological effectiveness of H3.3-K27M neoantigen vaccine for the treatment of DIPG patients | baseline 1: pre-radiotherapy; baseline 2: immediately after completing radiotherapy; Day 15, Day 57, Day 85 and every 8 weeks thereafter until up to 2 years after the first shot.
  Immunological effectiveness is measured by an IFN-γ ELISPOT assay as number of spot-forming cells in one million peripheral blood mononuclear cells.

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Zhang, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No